CLINICAL TRIAL: NCT00023283
Title: Counseling Conditions for Thrice Weekly Buprenorphine in a Primary Care Clinic
Brief Title: Counseling Conditions for Buprenorphine in a Primary Care Clinic - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Richard S. Schottenfeld, MD, Yale University School of Medicine
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: NIDA-9803-1; R01DA009803 (NIH); R01-9803-1
Record Dates: First submitted 2001-08-30; First posted 2001-08-31 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Heroin Dependence; Opioid-Related Disorders; Substance Abuse, Intravenous
Keywords: Opioid-Related Disorders
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders; Substance Abuse, Intravenous | interventions — Buprenorphine

ARMS (3):
- 1 (Experimental): Standard Medical Management with once-weekly medication dispensing
  Interventions: Drug: Buprenorphine
- 2 (Experimental): Standard Medical Management with thrice-weekly medication dispensing
  Interventions: Drug: Buprenorphine
- 3 (Experimental): Enhanced Medical Management with thrice-weekly medication dispensing
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — 1. Experimental Standard Medical Management with once-weekly medication dispensing
  2. Experimental Standard Medical Management with thrice-weekly medication dispensing
  3. Experimental Enhanced Medical Management with thrice-weekly medication dispensing

SUMMARY:
The purpose of this study is to compare the Standard Medical Management (SMM) vs. SMM enhanced with additional education about addiction and recovery (Enhanced Medical Management, EMM)

DETAILED DESCRIPTION:
A randomized trial, in a hospital primary care clinic, for 24 weeks, of 168 opioid-dependent subjects, maintained on buprenorphine 3x/week, and counseled with Standard or Enhanced Medical Management. SMM is a brief intervention similar to that provided by primary practitioners to patients with chronic medical conditions such as diabetes. EMM is an intervention that provides education about the recovery process and advice about lifestyle changes and 12-step participation. Outcome measures include reduction in opioid use and abstinence from opioids, documented by 3x/week urine testing and self report.

ELIGIBILITY:
Inclusion criteria: Subjects meeting FDA criteria for opioid agonist maintenance treatment and DSM-IV criteria for opioid dependence will be eligible for the study. Women of childbearing age will be included provided they agree to adequate contraception and to monthly pregnancy monitoring throughout the study.

Exclusion criteria include: pregnancy, current dependence on alcohol, benzodiazepines or sedatives; current suicide or homicide risk; current psychotic disorder or major depression; inability to read or understand English; life-threatening or unstable medical problems.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2000-08; Primary Completion 2003-12 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Self-reported frequency of illicit opioid use | 6 months
Percentage of opioid-negative urine specimens | 6 months
Maximum number of weeks abstinent from illicit opioids | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schottenfeld, M.D., Principal Investigator — Yale University
Locations (1):
- APT Residential Services Division, New Haven, Connecticut, United States

REFERENCES:
- [Derived] McHugh RK, Bailey AJ, McConaghy BA, Weiss RD, Fiellin DA, Hillhouse M, Moore BA, Fitzmaurice GM. Behavioral Therapy as an Adjunct to Buprenorphine Treatment for Opioid Use Disorder: A Secondary Analysis of 4 Randomized Clinical Trials. JAMA Netw Open. 2025 Aug 1;8(8):e2528529. doi: 10.1001/jamanetworkopen.2025.28529. PMID 40833692
- [Derived] Sullivan LE, Moore BA, Chawarski MC, Pantalon MV, Barry D, O'Connor PG, Schottenfeld RS, Fiellin DA. Buprenorphine/naloxone treatment in primary care is associated with decreased human immunodeficiency virus risk behaviors. J Subst Abuse Treat. 2008 Jul;35(1):87-92. doi: 10.1016/j.jsat.2007.08.004. Epub 2007 Oct 15. PMID 17933486
- [Derived] Fiellin DA, Pantalon MV, Chawarski MC, Moore BA, Sullivan LE, O'Connor PG, Schottenfeld RS. Counseling plus buprenorphine-naloxone maintenance therapy for opioid dependence. N Engl J Med. 2006 Jul 27;355(4):365-74. doi: 10.1056/NEJMoa055255. PMID 16870915